CLINICAL TRIAL: NCT02853097
Title: Studies of Cell-Free DNA and RNA in Blood From Patients Being Treated for Prostate Cancer
Brief Title: Cell-Free DNA and RNA in Blood fromMetastatic Prostate Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4P-15-4; NCI-2016-00958 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-15-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (blood collection): Patients undergo blood collection every 4-12 weeks during ADT, abiraterone, enzalutamide, or docetaxel treatment. Patients switched from ADT to either abiraterone or enzalutamide during the study will undergo phlebotomy every 6-12 weeks. Samples are analyzed for cfRNA, and cfDNA, AR-V7, and other AR-Vs via quantitative RT-PCR.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo blood collection
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies cell-free deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) in blood from patients with prostate cancer that does not respond to hormone therapy and has spread to other places in the body. Studying samples of blood from patients with prostate cancer may help doctors to learn more about the changes that occur in tumor cells over time and how they become resistant to anti-cancer drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To document the appearance of androgen receptor isoform splice variant 7 (AR-V7) expression over the course of therapy in castration-resistant prostate cancer (CRPC).

II. To determine whether detectable AR-V7 is associated with a shortened duration of treatment benefit of abiraterone or enzalutamide.

SECONDARY OBJECTIVES:

I. To determine how the presence and expression level of AR-V7 impacts response to docetaxel.

II. To determine at what point AR-V7 arises during androgen deprivation therapy (ADT) and how its presence and expression corresponds to castration resistance.

TERTIARY OBJECTIVES:

I. To determine if androgen receptor isoform splice variants (AR-Vs) other than AR-V7 play a role in resistance and / or response to the therapies explored in this study.

II. To determine if, in patients who do not express mutations in androgen receptor (AR), other genetic alterations are associated with treatment outcomes to the therapies explored in this study.

OUTLINE:

Patients undergo blood collection every 4-12 weeks during ADT, abiraterone and / or enzalutamide and docetaxel. Patients switched from ADT to either abiraterone or enzalutamide during the study will undergo phlebotomy every 6-12 weeks. Samples are analyzed for cell-free ribonucleic acid (cfRNA), cell-free deoxyribonucleic acid (cfDNA), AR-V7, and other AR-Vs via quantitative reverse transcriptase-polymerase chain reaction (RT-PCR).

After completion of study, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of histologically confirmed prostate adenocarcinoma and falling into one of the following 5 groups:

  * Currently receiving ADT (previously untreated for metastatic disease)

    * These patients will be grouped into 3 cohorts: having received ADT for 3-6 months; for 1-2 years; and for > 3 years
  * Scheduled to begin treatment with ADT (previously untreated for metastatic disease)
  * Scheduled to begin treatment with enzalutamide (castration resistant / has received ADT / may have received abiraterone)
  * Scheduled to begin treatment with abiraterone (castration resistant / has received ADT / may have received enzalutamide)
  * Scheduled to begin treatment with docetaxel (castration resistant / has received ADT / has received enzalutamide and/or abiraterone)
* Have been diagnosed with either hormone-naive or castrate-resistant metastatic disease
* Ability and willingness to provide written and informed consent

Exclusion Criteria:

* Patients who receive combined ADT with docetaxel for hormone-naive metastatic prostate cancer
* Patients on intermittent ADT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients at various points throughout androgen deprivation therapy and at the initiation of androgen deprivation therapy, enzalutamide, abiraterone and docetaxel with either computed tomography measurable or evaluable disease or arising prostate specific antigen disease
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2020-09-27 (Actual)

PRIMARY OUTCOMES:
Change in AR-V7 presence | Baseline to 3 years
  Each of the 4 longitudinal cohorts will be analyzed separately (at least initially). Kaplan-Meier-like curves (likely adjusted for interval censoring) will be used to display the development of AR-V7 positivity. To complement the analysis of Cohort A, an exact logistic regression analysis will be used with the data from Cohort X with AR-V7 splice variant positivity as the dependent variable and time since start of ADT as the independent variable. Logistic regression will be used to assess the association between AR-V7 status at start of treatment and overall response to treatment.
Expression level of AR-V7 in serum cfRNA assessed by quantitative RT-PCR | Up to 3 years
  Detectable AR-V7 will be associated with a shortened duration of treatment benefit (ADT, abiraterone, enzalutamide, docetaxel). Each of the 4 longitudinal cohorts will be analyzed separately (at least initially). A regression analysis based on the Cox proportional hazards model (if proportional hazards holds) will be used to assess the association between AR-V7 and time to new treatment. Initially, only the baseline AR-V7 status will be used. Next, AR-V7 will be included as a time dependent covariate; the model used may be modified to accommodate competing risks (if too many switch treatment p
Time to start of another treatment | Time from start of treatment until the time that the patient begins another therapy, assessed up to 3 years

SECONDARY OUTCOMES:
Expression levels of AR-Vs (other than AR-V7) in serum cfRNA assessed by quantitative RT-PCR | Up to 3 years
Tumor response as measured by Prostate Cancer Working Group | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, MD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California